CLINICAL TRIAL: NCT01543282
Title: Randomized Controlled Study Comparing Endoscopic Ultrasonography Guided Fine Needle Aspiration Using Free Stylet 22g and 25 g Needles in Solid Lesions
Brief Title: Endoscopic Ultrasonography (EUS) Guided Fine Needle Aspiration Using Free Stylet 22g and 25 g Needles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CE 11.150
Record Dates: First submitted 2011-12-15; First posted 2012-03-02 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Solid Neoplasms
Keywords: endoscopic ultrasonography; fine needle aspiration cytology; 22 gauge; 25 gauge

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EUS 22 gauge needle (Active Comparator): EUS 22 g needle is the most common needle used in clinical practice. EUS-FNA passes will be performed without stylet until sample adequacy or until a maximum of 5 FNA passes in pancreatic lesions or 3 FNA passes in other lesions. In case of inadequate sample after 3 passes, or needle failure, cross over to the other type of needle is allowed.
  Interventions: Device: Endosonography guided fine needle aspiration cytology ( Cook Medical, Boston Scientific)
- EUS 25 gauge needle (Experimental): 25 gauge needle is usually used less frequently but nowadays is increasingly used and is as well a valid option. EUS-FNA passes will be performed without stylet until sample adequacy or until a maximum of 5 FNA passes in pancreatic lesions or 3 FNA passes in other lesions. In case of inadequate sample after 3 passes, or needle failure, cross over to the other type of needle is allowed.
  Interventions: Device: Endosonography guided fine needle aspiration cytology ( Cook Medical, Boston Scientific)

INTERVENTIONS:
Device: Endosonography guided fine needle aspiration cytology ( Cook Medical, Boston Scientific) — Patients will be randomized either to receive EUS-FNA with a 22 g needle or 25 g needle. EUS-FNA passes will be performed without stylet until sample adequacy or until a maximum of 5 FNA passes in pancreatic lesions or 3 FNA passes in other lesions. In case of inadequate sample after 3 passes, or needle failure, cross over to the other type of needle is allowed.
  Other Names: Cook Medical; Boston Scientific

SUMMARY:
This is a randomized controlled study comparing EUS-FNA with 22 gauge and 25 gauge needles in consecutive patients.

Summary

Background: three needle sizes for endoscopic ultrasonography guided fine needle aspiration (EUS-FNA) are currently available: 22 Gauge (G), 25 G and 19 G. However, well design studies comparing them regarding efficacy and feasibility are lacking.

Aims: to investigate diagnostic yield, specimen adequacy, feasibility and complications of the conventional 22 G compared with the 25 G needle.

Methods: patients ≥ 18 years, referred to EUS-FNA for a solid lesion will be considered for inclusion. Patients with suspected diagnosis of lymphoma, GIST, sarcoidosis, significant coagulopathy (APT < 50% or platelets < 50000/mm3), use of warfarin or other anticoagulants, use of clopidogrel within 7 days of EUS, inability or refusal to sign the informed consent and pregnancy or suspected pregnancy will be excluded.

Participants will be randomized to 22 G needle and 25 G FNA. Chi-square test will be used to compare proportions. Continuous variables will be compared using Student´s t test. A two-tailed P values of less than 0.05 will be considered statistically significant. The diagnostic yield of 25 G and 22 G needle will be evaluated by four criteria: sensitivity, specificity, positive predictive value and negative predictive value. An expected rate of 85% diagnostic yield from EUS guided FNA by using 22G needle will be considered. By using a power of 80% and an α value of 0.05 would be necessary 120 patients per group to detect a 15% difference in the rate of diagnostic yield.

DETAILED DESCRIPTION:
1. Objectives

PRIMARY To compare diagnostic yield of stylet-free, solid lesion EUS-FNA using the 22 G FNA vs the 25 G FNA needle, in consecutive patients referred to EUS-FNA.

SECONDARY

To investigate:

1. specimen adequacy,
2. number of FNA passes,
3. ease of puncture,
4. failure of the FNA needle and
5. complications

3. Methods

3.1. Design: prospective randomized trial.

3.2. Inclusion: Consecutive patients referred for EUS-FNA of a solid lesion will be considered for inclusion.

3.3. Exclusion: Age < 18 years, patients with suspected diagnosis of lymphoma, GIST, sarcoidosis or other lesions in which a large amount of tissue will be required for diagnosis, significant coagulopathy (INR > 1.5, platelets < 50000/mm3, use of low molecular weight heparin, use of clopidogrel within 7 days of EUS), cystic lesions, or inability or refusal to sign the informed consent.

3.4. Endoscopic procedures: Informed consent will be obtained before each procedure by one of the researchers. Patients will not receive economic compensation or reimbursement of their expenses for coming to the exploration, since it is a procedure previously indicated. Then, potential candidates will be randomized to 22 G or 25 G FNA using a computer generated random sequence. There will be block randomization for a) pancreatic masses, 2) lymph nodes, or 3) all other lesions.

All examinations will be performed by two experienced endosonographers with a lineal echoendoscope (AS and SP). EUS procedures will be carried out with the patient, in left lateral position under conscious sedation using midazolam (2.5-5 mg) plus meperidine (50-100 mg) and droperidol (2.5-5 mg). Before performing the EUS-FNA biopsy, a complete examination of the pancreas, liver as well as other vicinity organs will be performed.

EUS-FNA passes will be performed without stylet until sample adequacy or until a maximum of 5 FNA passes in pancreatic lesions or 3 FNA passes in other lesions. In case of inadequate sample after 3 passes, or needle failure, cross over to the other type of needle is allowed. Ease of puncture will be scored qualitatively as poor (scored 1), good (scored 2) or excellent (scored 3).[14] FNA failure will be also reported. All procedures will be digitally videotaped. The examinations will be reviewed by a endosonographer blinded to the type of needle used and visibility of the needle will be scored (score 1 "poor", score 2 "good", score 3 "excellent").[14] After the procedure, patients will be monitored in the recovery room at least 60 minutes before discharge. Immediate complications will be assessed and recorded by nurses and/or physicians during and after the procedure while the patient was recovering from sedation.

3.5. Cytological analysis: All passes will be read by one experienced cytopathologist on-site utilizing microscopic evaluation of air-dried slides stained with Diff-Quik (International Reagents Co., Ltd., Kobe, Japan). The cytopathologist will be blinded to the type of needle used. The final cytological diagnosis was made using a standard Papanicolaou stain. For each lesion, the cytologist assessed sample adequacy: cellularity (score 1 "poor", score 2 "good", score 3 "excellent"),[14] and bloodiness (score 1 "minimal", score 2 "moderate", score 3 "significant")[21] and the presence or absence of malignancy ("positive"/"negative"/"suspicious"/ inconclusive).

3.6. Follow up Lesions will be considered malignant in the following cases: positive cytological diagnosis, positive histological diagnosis and clinical or radiological progression in the next 6 months. In case of negative results in the cytological diagnosis absence of clinical worsening and radiologic progression at least in the following 6 months after FNA will be required.

3.7. Data collection Clinical data will be prospectively collected and saved in a database including: demographic information (age and gender), size and location of the target lesion (pancreas, lymph node, liver, adrenal gland, others) and technical and procedure variables: FNA path (esophagus, stomach, duodenum), number of needle passes, needle visibility, ease to puncture, needle failure, cellularity, bloodiness, cytological diagnosis, final diagnosis, immediate complications.

4. Statistical analysis Results for continuous variables will be expressed as means and standard deviations. Categorical variables will be expressed as frequencies and percentages. Chi-square test will be used to compare proportions. Continuous variables will be compared using Student´s t test. A two-tailed P values of less than 0.05 will be considered statistically significant. Data were analyzed with the Statistical Package for Social Sciences v. 15.0 (SPSS Inc., Chicago, IL, USA). The diagnostic yield of 15 G and 22 G needle will be evaluated by four criteria: sensitivity, specificity, positive predictive value and negative predictive value.

Sample size An expected rate of diagnostic yield from EUS guided FNA by using 22G needle of 85% will be considered. By using a power of 80% and an α value of 0.05 would be necessary 120 patients per group to detect a 15% difference in the rate of diagnostic yield.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients referred for EUS-FNA of a solid lesion.

Exclusion Criteria:

* Age < 18 years
* Patients with suspected diagnosis of lymphoma, GIST, sarcoidosis or other lesions in which a large amount of tissue will be required for diagnosis
* Significant coagulopathy (INR > 1.5, platelets < 50000/mm3
* Use of low molecular weight heparin, use of clopidogrel within 7 days of EUS)
* Cystic lesions
* Inability or refusal to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-12-10 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of stylet-free, solid lesion EUS-FNA using the 22 G FNA vs the 25 G FNA needle, in consecutive patients referred to EUS-FNA. | 6 months

SECONDARY OUTCOMES:
Specimen adequacy, number of FNA passes, ease of puncture, failure of the FNA needle and complications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anand V Sahai, MD, Principal Investigator — Hopital Saint Luc (Centre Hopitalier de l´Université du Montreal) Montreal, Quebec, Canada
Locations (1):
- Hopital Saint Luc (Centre Hopitalier de l´Université du Montreal), Montreal, Quebec, Canada

REFERENCES:
- [Result] Yusuf TE, Ho S, Pavey DA, Michael H, Gress FG. Retrospective analysis of the utility of endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) in pancreatic masses, using a 22-gauge or 25-gauge needle system: a multicenter experience. Endoscopy. 2009 May;41(5):445-8. doi: 10.1055/s-0029-1214643. Epub 2009 May 5. PMID 19418399
- [Result] Imazu H, Uchiyama Y, Kakutani H, Ikeda K, Sumiyama K, Kaise M, Omar S, Ang TL, Tajiri H. A prospective comparison of EUS-guided FNA using 25-gauge and 22-gauge needles. Gastroenterol Res Pract. 2009;2009:546390. doi: 10.1155/2009/546390. Epub 2009 Nov 17. PMID 19997511
- [Result] Lee JH, Stewart J, Ross WA, Anandasabapathy S, Xiao L, Staerkel G. Blinded prospective comparison of the performance of 22-gauge and 25-gauge needles in endoscopic ultrasound-guided fine needle aspiration of the pancreas and peri-pancreatic lesions. Dig Dis Sci. 2009 Oct;54(10):2274-81. doi: 10.1007/s10620-009-0906-1. Epub 2009 Aug 11. PMID 19669880
- [Result] Sakamoto H, Kitano M, Komaki T, Noda K, Chikugo T, Dote K, Takeyama Y, Das K, Yamao K, Kudo M. Prospective comparative study of the EUS guided 25-gauge FNA needle with the 19-gauge Trucut needle and 22-gauge FNA needle in patients with solid pancreatic masses. J Gastroenterol Hepatol. 2009 Mar;24(3):384-90. doi: 10.1111/j.1440-1746.2008.05636.x. Epub 2008 Nov 20. PMID 19032453
- [Result] Camellini L, Carlinfante G, Azzolini F, Iori V, Cavina M, Sereni G, Decembrino F, Gallo C, Tamagnini I, Valli R, Piana S, Campari C, Gardini G, Sassatelli R. A randomized clinical trial comparing 22G and 25G needles in endoscopic ultrasound-guided fine-needle aspiration of solid lesions. Endoscopy. 2011 Aug;43(8):709-15. doi: 10.1055/s-0030-1256482. Epub 2011 May 24. PMID 21611946
- [Result] Fabbri C, Polifemo AM, Luigiano C, Cennamo V, Baccarini P, Collina G, Fornelli A, Macchia S, Zanini N, Jovine E, Fiscaletti M, Alibrandi A, D'Imperio N. Endoscopic ultrasound-guided fine needle aspiration with 22- and 25-gauge needles in solid pancreatic masses: a prospective comparative study with randomisation of needle sequence. Dig Liver Dis. 2011 Aug;43(8):647-52. doi: 10.1016/j.dld.2011.04.005. Epub 2011 May 17. PMID 21592873
- [Result] Wani S, Gupta N, Gaddam S, Singh V, Ulusarac O, Romanas M, Bansal A, Sharma P, Olyaee MS, Rastogi A. A comparative study of endoscopic ultrasound guided fine needle aspiration with and without a stylet. Dig Dis Sci. 2011 Aug;56(8):2409-14. doi: 10.1007/s10620-011-1608-z. Epub 2011 Feb 17. PMID 21327919